CLINICAL TRIAL: NCT03047265
Title: Phase II Randomized Trial Comparing Paclitaxel Combined With DDP Plus Concurrent Chemoradiotherapy With DDP Plus Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ling Guo, PROFESSOR, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 308-2016-02-01
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel (Experimental): Paclitaxel plus Cisplatin combine with IMRT
  Interventions: Drug: Paclitaxel
- Cisplatin (Active Comparator): Cisplatin combine with IMRT
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 135mg / m2 D1, DDP 20mg / m2 D1-4, D1,D29 of RT, a total of 2 courses.
  Other Names: TAXOL
  Arms: Paclitaxel
Drug: Cisplatin — Cisplatin 100mg / m2 , D1,D22,D43 of RT, a total of 3 courses.
  Other Names: DDP
  Arms: Cisplatin

SUMMARY:
This is a Phase II Randomized Trial to Compare Paclitaxel combined with DDP Plus Concurrent Chemoradiotherapy With DDP Plus Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma is one of the most common malignancies in South China. Nasopharyngeal carcinoma is sensitive to radiotherapy and chemotherapy. Concurrent chemoradiation has become a standard treatment for locally advanced stage III-IVb nasopharyngeal carcinoma. However, The recommended single-agent DDP concurrent chemotherapy regimen for high-risk patients (IVa-IVb period) to improve the efficacy was not significant. Paclitaxel combined with platinum in the same period of chemotherapy regimen has been widely used in head and neck cancer, cervical cancer, esophageal squamous cell carcinoma and lung cancer and other tumors, a number of studies have shown that it has good tolerance and efficacy. And a number of previous studies have shown that paclitaxel combined with platinum chemotherapy in the same period of head and neck cancer or nasopharyngeal cancer in multiple phase II clinical trials to achieve encouraging results. Based on the above background and basis, for the high risk (IVa-IVb) nasopharyngeal carcinoma treatment, the applicant intends to carry out the first IMRT + paclitaxel + DDP concurrent chemotherapy compared with DDP single drug concurrent chemotherapy regimen Pharyngeal cancer in a prospective randomized controlled phase Ⅱ clinical trial for paclitaxel + DDP dual-chemotherapy regimen for the treatment of high-risk nasopharyngeal carcinoma to provide evidence-based basis. (IVa-IVb) nasopharyngeal carcinoma (NPC), and to provide a high-level evidence-based evidence-based approach to the treatment of nasopharyngeal carcinoma at high risk (stage IVa-IVb). The results of this study will be used in international guidelines to optimize high- Treatment of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing carcinoma.
2. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III.
3. Original clinical staged as IVa-IVb（according to the 7th AJCC edition）.
4. Male and no pregnant female
5. Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1.
6. WBC ≥ 4×109 /L and PLT ≥4×109 /L and HGB ≥90 g/L
7. With normal liver function test (ALT、AST ≤ 2.5×ULN, TBIL≤ 2.0×ULN)
8. With normal renal function test (Creatinine ≤ 1.5×ULN)
9. Written informed consent.

Exclusion Criteria:

1. Patients have evidence of relapse or distant metastasis Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
2. Receiving radiotherapy or chemotherapy previously
3. The presence of uncontrolled life-threatening illness
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
5. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.

   Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
6. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
7. Concurrent systemic steroid therapy
8. HIV positive
9. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2017-02-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year progress free survival(PFS) | 3 years
  PFS means assignment to the date of any local or distant progress of the disease using Kaplan-Meier calculate the progress free survival rates,and find out is there significant difference between these two groups

SECONDARY OUTCOMES:
overall survival(OS) | 2 years ,3 years and 5 years
  the overall survival denote to assignment to date of death from any cause. Using Kaplan-Meier to calculate the 2-year ,3-year,5-year overall survival rate,and find is there any significant difference between these two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Langendijk JA, Leemans CR, Buter J, Berkhof J, Slotman BJ. The additional value of chemotherapy to radiotherapy in locally advanced nasopharyngeal carcinoma: a meta-analysis of the published literature. J Clin Oncol. 2004 Nov 15;22(22):4604-12. doi: 10.1200/JCO.2004.10.074. PMID 15542811
- [Background] Chen QY, Wen YF, Guo L, Liu H, Huang PY, Mo HY, Li NW, Xiang YQ, Luo DH, Qiu F, Sun R, Deng MQ, Chen MY, Hua YJ, Guo X, Cao KJ, Hong MH, Qian CN, Mai HQ. Concurrent chemoradiotherapy vs radiotherapy alone in stage II nasopharyngeal carcinoma: phase III randomized trial. J Natl Cancer Inst. 2011 Dec 7;103(23):1761-70. doi: 10.1093/jnci/djr432. Epub 2011 Nov 4. PMID 22056739
- [Background] Lin JC, Liang WM, Jan JS, Jiang RS, Lin AC. Another way to estimate outcome of advanced nasopharyngeal carcinoma--is concurrent chemoradiotherapy adequate? Int J Radiat Oncol Biol Phys. 2004 Sep 1;60(1):156-64. doi: 10.1016/j.ijrobp.2004.03.002. PMID 15337551
- [Background] Chen WH, Tang LQ, Guo SS, Chen QY, Zhang L, Liu LT, Qian CN, Guo X, Xie D, Zeng MS, Mai HQ. Prognostic Value of Plasma Epstein-Barr Virus DNA for Local and Regionally Advanced Nasopharyngeal Carcinoma Treated With Cisplatin-Based Concurrent Chemoradiotherapy in Intensity-Modulated Radiotherapy Era. Medicine (Baltimore). 2016 Feb;95(5):e2642. doi: 10.1097/MD.0000000000002642. PMID 26844482
- [Background] Garden AS, Harris J, Vokes EE, Forastiere AA, Ridge JA, Jones C, Horwitz EM, Glisson BS, Nabell L, Cooper JS, Demas W, Gore E. Preliminary results of Radiation Therapy Oncology Group 97-03: a randomized phase ii trial of concurrent radiation and chemotherapy for advanced squamous cell carcinomas of the head and neck. J Clin Oncol. 2004 Jul 15;22(14):2856-64. doi: 10.1200/JCO.2004.12.012. PMID 15254053